CLINICAL TRIAL: NCT01879826
Title: Efficacy of Laser Therapy as an Adjuvant Treatment During Kidney Biopsies to Decrease Anxiety and Pain.
Brief Title: Pediatric Laser Acupuncture and Renal Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Cynthia Kim, Associate Professor of Pediatrics, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Laser
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain; Anxiety
Keywords: Aculaser; Microlight ML830; Kidney biopsy; Pain; Anxiety; Sedation
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aculaser applied to sham points (Sham Comparator): The patient will receive aculaser, performed by licensed acupuncturist, to "sham" acupuncture sites. In addition, the patient will still receive standard pain control protocols with anesthetic medications like lidocaine plus ketamine or fentanyl and versed during the biopsy, along with pain management after the procedure.
  Interventions: Device: Aculaser applied to sham points
- Aculaser applied to kidney points (Experimental): The patient will receive aculaser, performed by licensed acupuncturist, to known kidney acupuncture sites. In addition, the patient will still receive standard pain control protocols with anesthetic medications like lidocaine plus ketamine or fentanyl and versed during the biopsy, along with pain management after the procedure.
  Interventions: Device: Aculaser applied to kidney points

INTERVENTIONS:
Device: Aculaser applied to kidney points — The patient will receive aculaser, performed by licensed acupuncturist, to known kidney acupuncture sites. In addition, the patient will still receive standard pain control protocols with anesthetic medications like lidocaine plus ketamine or fentanyl and versed during the biopsy, along with pain management after the procedure.
  Other Names: Aculaser: Microlight ML830
  Arms: Aculaser applied to kidney points
Device: Aculaser applied to sham points — The patient will receive aculaser, performed by licensed acupuncturist, to "sham" acupuncture sites. In addition, the patient will still receive standard pain control protocols with anesthetic medications like lidocaine plus ketamine or fentanyl and versed during the biopsy, along with pain management after the procedure.
  Other Names: Aculaser: Microlight ML830
  Arms: Aculaser applied to sham points

SUMMARY:
The purpose of this study is to test if treatment with laser therapy in pediatric patients undergoing renal biopsies will improve patient satisfaction of the overall procedure. In this study, the participant will receive a laser acupuncture treatment targeting either kidney acupoints or targeting "sham" points not associated with the kidney; the participant will not get both. Both treatment sessions are given by a certified medical acupuncturist. The patient will still receive standard pain control protocols with anesthetic medications like lidocaine plus ketamine or fentanyl and versed during the biopsy, along with pain management after the procedure. All medication will be administered without regard for which group the participant has been randomized, as the treatment team will also be blinded.

Hypothesis:

We will test the hypothesis that treatment with laser acupuncture in patients undergoing renal biopsies will improve patient satisfaction of the overall procedure.

Specific Aims:

Specific Aim 1: Determine whether the use of laser acupuncture improves patient's overall satisfaction of renal biopsy.

Specific Aim 2: Determine whether the use of laser acupuncture decreases the amount of sedative medication given during renal biopsy.

DETAILED DESCRIPTION:
At University of California San Francisco, there are approximately 100 pediatric renal biopsies per year. All of these patients receive sedation, which is prescribed and supervised by the pediatric pain and palliative care team, with either ketamine or fentanyl and versed. Child life is involved; however, many children still experience anxiety and/or pain with the procedure. Use of a modality such as aculaser which may decrease these symptoms could enhance their experience.

The term "laser" stands for light amplification by stimulated emission of radiation. In laser acupuncture, a low power, cold light produced by a low-level laser diode is used to stimulate an acupuncture point. As it is non-invasive, laser acupuncture is thought to be safer than needle acupuncture, especially in the setting of patients with blood-borne infectious diseases. In a systematic review analyzing the evidence to support the effectiveness of laser acupuncture, randomized control trials in which adults with soft tissue injury, acute or chronic pain condition, or any systemic illness were included. This review reports moderate level of evidence for treatment of myofascial pain and post-operative nausea/vomiting and limited evidence of the clinical effectiveness of treating chronic tension headaches. Of note, no complications of the use of aculaser were reported in this review (1).

1. Baxter GD, Bleakley C, McDonough S. Clinical effectiveness of laser acupuncture: a systematic review. J Acupunct Meridian Stud. 2008 Dec;1(2):65-82.

ELIGIBILITY:
Inclusion Criteria:

* older than 6 years old
* admitted for a transplant or native kidney biopsy performed by pediatric nephrology

Exclusion Criteria:

* Prisoners
* Pregnant females
* Those who are unable to participate with the visual analog scale

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Kim, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Baxter GD, Bleakley C, McDonough S. Clinical effectiveness of laser acupuncture: a systematic review. J Acupunct Meridian Stud. 2008 Dec;1(2):65-82. doi: 10.1016/S2005-2901(09)60026-1. PMID 20633458
- [Result] Schlager A, Offer T, Baldissera I. Laser stimulation of acupuncture point P6 reduces postoperative vomiting in children undergoing strabismus surgery. Br J Anaesth. 1998 Oct;81(4):529-32. doi: 10.1093/bja/81.4.529. PMID 9924226
- [Result] Gottschling S, Meyer S, Gribova I, Distler L, Berrang J, Gortner L, Graf N, Shamdeen GM. Laser acupuncture in children with headache: a double-blind, randomized, bicenter, placebo-controlled trial. Pain. 2008 Jul 15;137(2):405-412. doi: 10.1016/j.pain.2007.10.004. Epub 2007 Nov 19. PMID 18022318
- [Result] Resim S, Gumusalan Y, Ekerbicer HC, Sahin MA, Sahinkanat T. Effectiveness of electro-acupuncture compared to sedo-analgesics in relieving pain during shockwave lithotripsy. Urol Res. 2005 Aug;33(4):285-90. doi: 10.1007/s00240-005-0473-7. Epub 2005 Jun 22. PMID 15971087
- [Derived] Oates A, Benedict KA, Sun K, Brakeman PR, Lim J, Kim C. Laser acupuncture reduces pain in pediatric kidney biopsies: a randomized controlled trial. Pain. 2017 Jan;158(1):103-109. doi: 10.1097/j.pain.0000000000000734. PMID 27749608

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aculaser Applied to Sham Points | Aculaser Applied to Kidney Points
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aculaser Applied to Sham Points | Aculaser Applied to Kidney Points | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Customized [Number; unit: participants]
  7-25 years | 41 | 40 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain/Anxiety
Description: The patient will complete a visual analog scale (rate 0-10) to assess pain after the procedure. Zero is no pain and 10 is worse pain. Change was calculated by baseline minus day one.
Time Frame: 1 day
Population: Number of participants in the final analysis were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aculaser Applied to Sham Points | Aculaser Applied to Kidney Points
Number analyzed (Participants) | 36 | 33
units on a scale | -0.5 (0.5) | 0.8 (0.4)
Statistical Analysis 1: Comparison: Aculaser Applied to Sham Points vs Aculaser Applied to Kidney Points; Test type: Non-Inferiority or Equivalence — With a power of 0.8 and an acceptable type I error size of 0.05, 38 patients per group was estimated to achieve significance; p = 0.044, t-test, 2 sided

2. Secondary Outcome: Parent Perception of Patient Pain Report
Description: Parent Perception of Patient Pain, scale is from 0 to 10, minimum value is 0, maximum value is 10, higher scores mean better outcome.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aculaser Applied to Sham Points | Aculaser Applied to Kidney Points
Number analyzed (Participants) | 36 | 33
units on a scale | 0.3 (0.5) | 2.3 (0.8)
Statistical Analysis 1: Comparison: Aculaser Applied to Sham Points vs Aculaser Applied to Kidney Points; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Aculaser Applied to Sham Points | Aculaser Applied to Kidney Points
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes